CLINICAL TRIAL: NCT00392301
Title: Split-Thickness Skin Graft Donor Site Wound Healing Study
Status: Withdrawn | Type: Observational
Why Stopped: Not funded - and PI left for another position in 2012
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Annette Wysocki, PhD, RN, Associate Dean for Research and Professor, University of Massachusetts, Amherst
Other Study IDs: 2006-0094
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Split-thickness Skin Graft Donor Sites
Keywords: wound healing; skin; graft donor site; donor site; transepidermal water loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to discover whether instruments widely used in skin research can be used to measure wound healing in split thickness skin graft donor sites and whether these instruments can detect differences in healing when two different dressing products are used.

DETAILED DESCRIPTION:
Currently there is no standard treatment to promote wound healing for split thickness skin graft donor sites and healing is determined based on clinical observation of the graft donor site and clinical judgement. Here we propose to use two instruments commonly used in skin research to measure wound healing. This study will validate the use of these two instruments, one that measures transepidermal water loss and the other that measures skin pigmentation to determine healing. To further validate the use of these instruments we will determine if these instruments can detect differences between two different wound dressing products that have been previously reported to heal skin graft donor sites at different rates.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age and over who have a split-thickness skin graft donor site.

Exclusion Criteria:

* Individuals under 18 years of age.
* Individuals who do not have a split thickness skin graft donor site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with split thickness skin graft donor sites
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10 (Estimated); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annette B. Wysocki, PhD, RN, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Disa JJ, Alizadeh K, Smith JW, Hu Q, Cordeiro PG. Evaluation of a combined calcium sodium alginate and bio-occlusive membrane dressing in the management of split-thickness skin graft donor sites. Ann Plast Surg. 2001 Apr;46(4):405-8. doi: 10.1097/00000637-200104000-00009. PMID 11324883
- [Background] Feldman DL, Rogers A, Karpinski RH. A prospective trial comparing Biobrane, Duoderm and xeroform for skin graft donor sites. Surg Gynecol Obstet. 1991 Jul;173(1):1-5. PMID 1907769
- [Background] Feldman DL. Which dressing for split-thickness skin graft donor sites? Ann Plast Surg. 1991 Sep;27(3):288-91. doi: 10.1097/00000637-199109000-00017. PMID 1952757
- [Background] Kilinc H, Sensoz O, Ozdemir R, Unlu RE, Baran C. Which dressing for split-thickness skin graft donor sites? Ann Plast Surg. 2001 Apr;46(4):409-14. doi: 10.1097/00000637-200104000-00010. PMID 11324884
- [Background] Malpass KG, Snelling CF, Tron V. Comparison of donor-site healing under Xeroform and Jelonet dressings: unexpected findings. Plast Reconstr Surg. 2003 Aug;112(2):430-9. doi: 10.1097/01.PRS.0000070408.33700.C7. PMID 12900600
- [Background] Rakel BA, Bermel MA, Abbott LI, Baumler SK, Burger MR, Dawson CJ, Heinle JA, Ocheltree IM. Split-thickness skin graft donor site care: a quantitative synthesis of the research. Appl Nurs Res. 1998 Nov;11(4):174-82. doi: 10.1016/s0897-1897(98)80296-6. PMID 9852660